CLINICAL TRIAL: NCT03138863
Title: Fetal Endoscopic Tracheal Occlusion (FETO) in Severe Left Congenital Diaphragmatic Hernia (CDH) NCT3138863
Brief Title: Fetal Endoscopic Tracheal Occlusion for Congenital Diaphragmatic Hernia (FETO)
Acronym: FETO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rodrigo Ruano (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Ruano, Professor and Chief of MFM Division, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220033-1; 16-008720 (Other: Mayo Clinic); NCT05339152 (obsolete NCT alias)
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Congenital Diaphragmatic Hernia; Pulmonary Hypoplasia; Pulmonary Artery Hypertension
Keywords: fetal lungs; fetal surgery; congenital diaphragmatic hernia; tracheal occlusion; pulmonary hypoplasia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- FETO Group (Experimental): Participants undergoing fetal endoscopic tracheal occlusion (FETO) surgery by insertion of the BALT GoldbBAL2 Detachable Balloon with the BALT catheter system.
  Interventions: Device: BALT GoldbBAL2 Detachable Balloon; Device: Catheter System

INTERVENTIONS:
Device: BALT GoldbBAL2 Detachable Balloon — Latex balloon, with radio-opaque inclusion
Device: Catheter System — 100 cm tapered micro-catheter
  Other Names: BALTACCIBDPE100

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of a new procedure called Fetoscopic Endoluminal Tracheal Occlusion (FETO).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Normal fetal karyotype with confirmation by culture results. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is > 26 weeks.
* Isolated Left CDH with liver up
* Gestation age at enrollment prior to 29 wks plus 6 days severe pulmonary hypoplasia with ultrasound (US) O/E lung area to head circumference ratio (LHR) < 25% (measured at 180 to 296 weeks) at the time of surgery; O/E LHR 25% to <30% (measured at 300 to 316 weeks) at time of surgery.
* Gestational age at FETO procedure with O/E LHR <25% at 27 weeks 0 days to 29 weeks 6 days; with O/E LHR 25% to <30% at 30 weeks 0 days to 31 weeks 6 days as determined by clinical information (LMP) and evaluation of first ultrasound
* Patient meets psychosocial criteria

Exclusion Criteria:

* Multi-fetal pregnancy
* History of natural rubber latex allergy
* Preterm labor, cervix shortened (<15 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
* Psychosocial ineligibility, precluding consent:
* Inability to reside within 30 minute drive of our hospital, and inability to comply with the travel for the follow-up requirements of the trial
* Patient does not have a support person (e.g. spouse, partner, mother) available to stay with the patient for the duration of the pregnancy at our institution.
* Right sided CDH or bilateral CDH, isolated left sided with O/E LHR ≥30% (measured at 180 to 295 weeks) as determined by ultrasound
* Additional fetal anomaly and chromosomal abnormalities by ultrasound, MRI, or echocardiogram at the fetal treatment center. No cases will be removed post hoc if abnormalities are discovered in the course of postoperative monitoring
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accrete) known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of successfully completed FETO procedures | Up to 34 weeks gestation
  The number of successful placement and removal of balloon during FETO procedure
Operative time | Up to 34 weeks gestation
  FETO placement and release operative times reported in minutes
Frequency of unplanned balloon removal | Up to 34 weeks gestation
  The frequency of non-emergent and emergent completion of FETO release (unplanned balloon removal)
Number of incidences of maternal complications | Up to 41 weeks gestation
  Maternal complications including preterm labor, premature rupture of membranes, oligohydramnios, polyhydramnios, chorioamnionitis
Number of participants with maternal complications | Up to 41 weeks gestation
  Maternal complications including preterm labor, premature rupture of membranes, oligohydramnios, polyhydramnios, chorioamnionitis
Gestational Age at Delivery | Up to 41 weeks gestation
  Gestation Age reported at time of delivery

SECONDARY OUTCOMES:
Fetal Lung Growth as measured via Fetal Lung Volume | Up to 41 weeks gestation
  Fetal Lung Volume as measured via ultrasound
Fetal Lung Growth as measured via LHR | Up to 41 weeks gestation
  Lung area to head circumference Ratio (LHR) as measured via ultrasound
Fetal survival | Up to 24 months post partum
  Fetal survival reported in days
Number of newborns reported at each oxygen dependency grading | Up to 24 months post partum
  Oxygen dependency graded as none, mild, moderate, severe as assessed by treating physician
Number of occurrence of severe pulmonary hypertension | Up to 24 months post partum
  Number of occurrence of severe pulmonary hypertension in infants as measured via echocardiogram
Number of infants requiring ECMO Support | Up to 24 months post partum
  Number of infants reported that required Extracorporeal membrane oxygenation (ECMO) support
Number of days in neonatal intensive care unit | Up to 24 months post partum
  Number of days infant was in the neonatal intensive care unit
Number of days of ventilator support | Up to 24 months post partum
  Number of reported days infants required ventilator support
Number of days of maternal hospitalization | Up to 24 months post partum
  Number of reported days of maternal hospitalization
Number of infants reporting presence of complications | Up to 24 months post partum
  Number of infants reporting the presence of: periventricular leucomalacia at < 2 months postnatally, neonatal sepsis, intraventricular hemorrhage (grade 0-III), retinopathy of prematurity (grade III or higher), gastro-esophageal reflux, tracheomegaly and tracheomalacia
Number of infants requiring the use of patch or muscle flap | Up to 24 months post partum
  Number of infants reported to require the use of patch or muscle flap
Number of participants at each route of delivery | Day 1 (post partum)
  Number of participants that delivered vaginally and via caesarean section
Number of days of Diaphragmatic Repair | Up to 24 months post partum
  Number of days of infant Diaphragmatic Repair

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruano, M.D., Ph.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No